CLINICAL TRIAL: NCT00626249
Title: A Phase 1b, Single-Dose, Open Label, Parallel Design, Controlled Pharmacology Trial of Fumaryl Diketopiperazine Administered as Technosphere Inhalation Power in Subjects With Either Mild or Moderate Chronic Kidney Disease vs. Matched Subjects Without Chronic Kidney Disease
Brief Title: Single Dose, Single Administration Study of Technosphere Inhalation Powder in Diabetic Subjects With Mild or Moderate Kidney Disease Compared to Diabetic Subjects With Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-T-017
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Mild Nephropathy; Moderate Nephropathy; Diabetes Mellitus
Keywords: Nephropathy; Kidney Disease; Diabetic; Renal; Diabetics
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases

ARMS (2):
- T Inhalation powder in diabetic subjs w/ normal renal func (Experimental): T inhalation powder in diabetic subjects with normal renal function, Single dose, 30 units
  Interventions: Drug: Technosphere Inhalation Powder
- T Inhalation powder diabetic subj w/mild or moderate nephrop (Experimental): T Inhalation powder in diabetic subjects w/mild or moderate nephropathy - Single dose, 30 units
  Interventions: Drug: Technosphere Inhalation Powder

INTERVENTIONS:
Drug: Technosphere Inhalation Powder — Technosphere Inhalation Powder

SUMMARY:
24 diabetics with mild & moderate renal disease and 12 diabetics without renal disease. One screening, one dosing & one follow-up visit with TechnosphereÂ® Inhalation Powder given at Visit 2 via MedToneÂ® Inhaler and PK testing at 26 designated time points

DETAILED DESCRIPTION:
This Phase 1, single-dose trial is being conducted to determine if nephropathy affects the way the kidneys eliminate the byproducts of TechnosphereÂ® Inhalation Powder as compared to kidneys free of disease. This trial will test the safety, tolerability and pharmacokinetics of the study medication. The trial consists of a screening, dosing and a follow-up visit. Single dose administration of TechnosphereÂ® Inhalation Powder occurs at the dosing visit. (V2) with serum and urine PK testing .

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking males and females, = 18 and = 80 years with a BMI of = 37 kg/m2
* Type 1 or type 2 diabetic
* Subjects with mild or moderate DNP and subjects with normal renal function, based on GFR rate and albuminuria
* Normal pulmonary function and performance based on PFTs

Exclusion Criteria:

* No history of COPD, asthma, or active respiratory infection; must be able to perform PFTs
* No dose and/or formulation changes within the preceding 6 weeks for any concomitant medications
* No clinically significant major organ/systemic disease
* No previous or current chemotherapy or radiation therapy that may result in pulmonary toxicity
* No clinically significant abnormalities on screening laboratory evaluation, except abnormal laboratory renal parameters in subjects with DNP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Differences in exposure to fumaryl diketopiperazine (FDKP) | 14 days

SECONDARY OUTCOMES:
Additional safety parameters | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Anders Boss, Study Director — Mannkind Corporation
Locations (3):
- United States (3):
  - Davita Clinical Research, Minneapolis, Minnesota
  - Qualia Clinical Research, Omaha, Nebraska
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas